CLINICAL TRIAL: NCT05953142
Title: Use of Dobutamine in Patients With Sepsis and Maintained Hypoperfusion After Initial Volemic Resuscitation.
Acronym: DEEP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Flavia Ribeiro Machado, Federal University of São Paulo, Federal University of São Paulo
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEEP
Record Dates: First submitted 2023-07-12; First posted 2023-07-19 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Sepsis; Hypoperfusion; Hyperlactatemia
Keywords: sepsis; hypoperfusion; dobutamine
MeSH Terms: conditions — Sepsis; Hyperlactatemia | interventions — Dobutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Patients in this group will receive the usual treatment according to the Surviving Sepsis Campaign guidelines.
- Dobutamine (Experimental): Patients in this group will receive, in addition to usual care, dobutamine in continuous infusion for a period of 48 hours after the randomization.
  Interventions: Drug: Dobutamine

INTERVENTIONS:
Drug: Dobutamine — Intravenous infusion of dobutamine in incremental dosis according to perfusion markers for a period of 48 hours after randomization.
  Arms: Dobutamine

SUMMARY:
This phase 2 study aim to investigate the effect of dobutamine in patients with sepsis/ septic shock after fluid resuscitation and with hypoperfusion (lactate and central venous oxygen saturation or prolonged capillary refill time) on renal function as compared with usual care.

DETAILED DESCRIPTION:
In this phase 2 study patients with sepsis/ septic shock and signs of persistent hypoperfusion after fluid resuscitation will be randomized to receive either dobutamine or no intervention in addition to usual care. Dobutamine will be used for 48 hours. Hypoperfusion will be assessed by altered lactate levels and a low SvO2 or prolonged capillary refill time. Both arms will receive usual care according to the Surviving Sepsis Campaign guidelines. Dobutamine dosis will be adjusted to achieve improvement in the perfusion parameters according to a pre specified protocol. Pre specified criteria will be used to stop the drug for safety. The primary outcome will be creatinine at Day 3. Other secondary and safety outcomes will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Patient with sepsis (suspected or confirmed) for less than 48 hours with:

Adequate volume resuscitation with 30 ml/kg of crystalloid solution or assessment by the attending physician that fluid resuscitation is no longer indicated Signs of hypoperfusion for less than 12 hours assessed by arterial lactate over two times the reference value and central venous saturation (SvcO2) less than 66% OR capillary refill time greater than 3 seconds.

Exclusion Criteria:

* Pregnancy
* Risk of imminent death within the next 12 hours in the opinion of the attending physician
* Patients under end of live care
* Previous congestive heart failure in functional class IV and/or dependence for all basic activities of daily living
* Hemoglobin levels below 7.0 g/dL
* Current use of dobutamine
* Patients in renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Serum creatine on the third day | 3 days
  Serum creatinine corrected by fluid balance on the third day

SECONDARY OUTCOMES:
ICU mortality | 60 days
  death in the ICU truncated at 60 days
Renal replacement therapy up to day 7 | 7 days
  need for renal replacement therapy within the first 7 days after randomization
Hospital mortality | 60 days
  death in the hospital truncated at 60 days
Vasopressors free days up to day 7 | 7 days
  Days without vasopressors support within the first 7days after randomization
ICU free days up to day 28th | 28 days
  Days out of the ICU within the first 28 days after randomization
Severe arrhythmia | 7 days
  Occurence of severe arrhythmia defined by the need for cardioversion (electric or chemical)

CONTACTS AND LOCATIONS:
Overall Officials: Amalia Pinguello, MD, Principal Investigator — Federal University of São Paulo; Flavia Machado, PhD, MD, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
unidentified patients data can be provided upon requested.